CLINICAL TRIAL: NCT00982007
Title: A Multi-center, Randomized, Active Controlled Study to Investigate the Efficacy and Safety of Intravenous Ferric Carboxymaltose (FCM) in Patients With Iron Deficiency Anemia (IDA)
Brief Title: Efficacy and Safety of Intravenous Ferric Carboxymaltose (FCM) in Patients With Iron Deficiency Anemia (IDA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT09031
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Iron Deficiency Anemia
Keywords: IDA
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Iron-Dextran Complex; ferryl iron; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Group A) - Ferric Carboxymaltose (FCM) (Experimental): Intravenous (IV) iron
  Interventions: Drug: Ferric Carboxymaltose (FCM)
- Cohort 1 (Group B) - Ferrous Sulfate (Active Comparator): Oral iron - Ferrous Sulfate tablets
  Interventions: Drug: Ferrous Sulfate Tablets
- Cohort 2 (Group D) - IV Iron (standard of care) (Active Comparator): Other IV iron
  Interventions: Drug: IV Iron (standard of care)
- Cohort 2 (Group C) - Ferric Carboxymaltose (FCM) (Experimental): Intravenous (IV) iron
  Interventions: Drug: Ferric Carboxymaltose (FCM)

INTERVENTIONS:
Drug: Ferric Carboxymaltose (FCM) — A total maximum cumulative dose of 1500 mg administered on Days 0 and 7.
  Arms: Cohort 1 (Group A) - Ferric Carboxymaltose (FCM)
Drug: Ferrous Sulfate Tablets — 325 mg Ferrous Sulfate tablets taken orally three times a day
  Arms: Cohort 1 (Group B) - Ferrous Sulfate
Drug: IV Iron (standard of care) — IV standard of care (other IV iron) per the Investigator's discretion
  Arms: Cohort 2 (Group D) - IV Iron (standard of care)
Drug: Ferric Carboxymaltose (FCM) — A total maximum cumulative dose of 1500 mg administered on Days 0 and 7.
  Arms: Cohort 2 (Group C) - Ferric Carboxymaltose (FCM)

SUMMARY:
The main objective of this study is to demonstrate the efficacy and safety of an investigational intravenous (IV) iron, ferric carboxymaltose (FCM), compared to oral iron in subjects who have iron deficiency anemia (IDA) and have shown an unsatisfactory response to oral iron.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ to 18 years of age and able to give informed consent.
* Diagnosis of Iron Deficiency Anemia (IDA).
* Hemoglobin (Hgb) ≤ to 11 g/dL.
* Ferritin ≤ to 100 ng/mL or ≤ 300 when Transferrin Saturation (TSAT) was ≤ 30%.
* Must demonstrate an unsatisfactory response or intolerance to oral iron.

Exclusion Criteria:

* Known hypersensitivity reaction to any component of ferric carboxymaltose or ferrous sulfate.
* Previously randomized in a clinical study of Ferric Carboxymaltose (FCM).
* Requires dialysis for treatment of chronic kidney disease.
* No evidence of iron deficiency.
* Any non-viral infection.
* AST or ALT at screen 1, as determined by central labs, greater than 1.5 times the upper limit of normal.
* Known positive hepatitis with evidence of active disease.
* Received an investigational drug within 30 days of screening.
* Alcohol or drug abuse within the past 6 months.
* Hemochromatosis or other iron storage disorders.
* Estimated life expectancy of less than 6 months or, for cancer patients, an ECOG Performance Status greater than 1.
* Any other laboratory abnormality, medical condition, or psychiatric disorders which in the opinion of the investigator would put the subject's disease management at risk or may result in the subject being unable to comply with study requirements.
* Pregnant or sexually-active females who are of childbearing potential and who are not willing to use an acceptable form of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 997 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals, Inc., Norristown, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals and Medical Clinics
Groups:
- Cohort 1 (Group A) - Ferric Carboxymaltose (FCM); Cohort 2 (Group C) - Ferric Carboxymaltose (FCM): Intravenous (IV) iron
  Ferric Carboxymaltose (FCM) : A total maximum cumulative dose of 1500 mg administered on Days 0 and 7.
- Cohort 1 (Group B) - Ferrous Sulfate: Oral iron
  Ferrous Sulfate Tablets : 325 mg Ferrous Sulfate tablets taken orally three times a day
- Cohort 2 (Group D) - IV Iron (Standard of Care): Other IV iron
  IV Iron (standard of care) : IV standard of care (other IV iron) per the Investigator's discretion
Period: Overall Study
Arm/Group | Cohort 1 (Group A) - Ferric Carboxymaltose (FCM) | Cohort 1 (Group B) - Ferrous Sulfate | Cohort 2 (Group C) - Ferric Carboxymaltose (FCM) | Cohort 2 (Group D) - IV Iron (Standard of Care)
Started | 250 | 257 | 253 | 251
Completed | 246 | 253 | 253 | 245
Not Completed | 4 | 4 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Group A) - Ferric Carboxymaltose (FCM) | Cohort 1 (Group B) - Ferrous Sulfate | Cohort 2 (Group C) - Ferric Carboxymaltose (FCM) | Cohort 2 (Group D) - IV Iron (Standard of Care) | Total
Number analyzed (Participants) | 246 | 253 | 253 | 245 | 997
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 7 | 2 | 3 | 14
  Between 18 and 65 years | 209 | 208 | 216 | 218 | 851
  >=65 years | 35 | 38 | 35 | 24 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (17.18) | 43.5 (17.71) | 43.6 (16.88) | 42.6 (15.51) | 43.2 (16.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233 | 238 | 239 | 231 | 941
  Male | 13 | 15 | 14 | 14 | 56
Region of Enrollment [Number; unit: participants]
  United States | 246 | 253 | 253 | 245 | 997

OUTCOME MEASURES:

1. Primary Outcome: Mean Increase From Baseline to the Highest Observed Hemoglobin Value Between Baseline and Day 35 or Time of Intervention for Patients Taking FCM as Compared to That for Patients Taking Ferrous Sulfate.
Time Frame: Day 35
Population: Modified Intent-to-Treat Population: Subjects who have received at least 1 dose of randomized study medication and had at least 1 post-baseline hemoglobin assessment
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Cohort 1 (Group A) - Ferric Carboxymaltose (FCM) | Cohort 1 (Group B) - Ferrous Sulfate | Cohort 2 (Group C) - Ferric Carboxymaltose (FCM) | Cohort 2 (Group D) - IV Iron (Standard of Care)
Number analyzed (Participants) | 244 | 251 | 245 | 237
g/dL | 1.57 (1.194) | 0.80 (0.799) | 2.90 (1.640) | 2.16 (1.252)

ADVERSE EVENTS:
Time Frame: 1 year and 6 months
Arm/Group | Cohort 1 (Group A) - Ferric Carboxymaltose (FCM) | Cohort 1 (Group B) - Ferrous Sulfate | Cohort 2 (Group C) - Ferric Carboxymaltose (FCM) | Cohort 2 (Group D) - IV Iron (Standard of Care)
Serious Adverse Events (participants affected / at risk) | 8/246 | 10/253 | 17/253 | 16/245
Other Adverse Events (participants affected / at risk) | 31/246 | 5/253 | 26/253 | 10/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Group A) - Ferric Carboxymaltose (FCM) (N=246) | Cohort 1 (Group B) - Ferrous Sulfate (N=253) | Cohort 2 (Group C) - Ferric Carboxymaltose (FCM) (N=253) | Cohort 2 (Group D) - IV Iron (Standard of Care) (N=245)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cystic fibrosis (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 3
Bacteremia (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Mastitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 2 | 2
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Uterine hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Group A) - Ferric Carboxymaltose (FCM) (N=246) | Cohort 1 (Group B) - Ferrous Sulfate (N=253) | Cohort 2 (Group C) - Ferric Carboxymaltose (FCM) (N=253) | Cohort 2 (Group D) - IV Iron (Standard of Care) (N=245)
Nausea (Gastrointestinal disorders) | 20 | 5 | 10 | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 11 | 0 | 16 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less